CLINICAL TRIAL: NCT06535607
Title: A Phase II, Multi-Center Study to Evaluate the Efficacy and Safety of Volrustomig as Monotherapy or in Combination With Anti-cancer Agents in Participants With Advanced/Metastatic Solid Tumors
Brief Title: Study of Volrustomig as Monotherapy or in Combination With Anti- Cancer Agents in Participants With Advanced/Metastatic Solid Tumors
Acronym: eVOLVE-02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D798MC00002
Record Dates: First submitted 2024-07-31; First posted 2024-08-02 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Cervical Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: cervical cancer; head and neck squamous cell carcinoma; eVOLVE-02; Volrustomig
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sub-study 1 (Experimental): Volrustomig monotherapy
  Interventions: Biological: Volrustomig
- Sub-study 2 (Experimental): Volrustomig monotherapy
  Interventions: Biological: Volrustomig
- Sub-study 3 (Experimental): Volrustomig in combination with carboplatin plus paclitaxel or 5-FU plus platinum
  Interventions: Biological: Volrustomig; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: Volrustomig — IV Infusion
Drug: Cisplatin — IV Infusion
  Arms: Sub-study 3
Drug: Carboplatin — IV Infusion
  Arms: Sub-study 3
Drug: Paclitaxel — IV Infusion
  Arms: Sub-study 3

SUMMARY:
eVOLVE-02 study will evaluate the efficacy and safety of volrustomig as monotherapy or in combination with anti-cancer agents in participants with advanced/metastatic solid tumors.

DETAILED DESCRIPTION:
eVOLVE-02 study will evaluate volrustomig monotherapy or volrustomig-based combination therapy in various advanced or metastatic solid tumors.

In sub-study 1, volrustomig will be evaluated as monotherapy in approximately 30 evaluable participants with cervical cancer.

In sub-study 2, volrustomig will be evaluated as monotherapy in approximately 20 evaluable participants with head and neck squamous cell carcinoma.

In sub-study 3, Volrustomig in Combination with Chemotherapy will be evaluated in approximately 60 evaluable participants with head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

1. Age ≥18 at the time of signing the ICF.
2. Provision of tumor sample to assess the PD-L1 expression.
3. Measurable disease according to RECIST 1.1.
4. ECOG performance status of 0 or 1.
5. Life expectancy ≥ 12 weeks.
6. Adequate organ and bone marrow function.
7. Body weight > 35 kg.
8. Capable of giving signed informed consent.
9. For sub-study 1, participants with R/M cervical cancer with squamous cell, adenocarcinoma or adenosquamous histology, that: have experienced disease progression during or after treatment with standard systematic therapy per local guideline; have received at least 1 line but no more than 2 lines of prior systemic treatment regimens for R/M cervical cancer.
10. For sub-study 2, for participants with OPC must have documented HPV status.
11. For sub-study 2, participants with R/M HNSCC, that: (a) Are histologically or cytologically documented R/M HNSCC of the OP, OC, HP, and LX that is considered incurable by local therapies; (b) Participants that have not been treated in R/M setting must have: (i) a documented PD-L1 positive result, (ii) with no prior systemic anti-cancer therapy for R/M HNSCC; (c) Platinum refractory participants must have relapsed from or are refractory to the first line of prior platinum-containing regimen.
12. For sub-study 3, participants with R/M HNSCC, that: (a) Are histologically or cytologically documented R/M HNSCC of the OP, OC, HP, and LX that is considered incurable by local therapies; (b) Participants that have not been treated in R/M setting

Exclusion Criteria

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Spinal cord compression.
2. Brain metastases unless asymptomatic, stable, and not requiring steroids for at least 14 days prior to start of study intervention.
3. Participants with primary neuroendocrine, mesenchymal, sarcomatoid histologies, or other histologies not mentioned as part of the inclusion criteria.
4. Have not recovered (ie, ≤ Grade 1 or at baseline) from an AE due to a previously administered anti-cancer therapy.
5. For sub-study 2, have had radiotherapy within 2 weeks prior to enrollment.
6. For sub-study 3, Participants have contraindications to any of the following drugs: 5-FU, paclitaxel and carboplatin
7. History of another primary malignancy except for a) Malignancy treated with curative intent with no known active disease ≥2 years before the first dose of study intervention and of low potential risk for recurrence; b) Adequately treated nonmelanoma skin cancer or lentigo maligna, or carcinoma in situ without evidence of disease.
8. Any evidence of diseases, and/or history of organ transplant or allogenic stem cell transplant, which makes it undesirable for the participant to participate in the study or that would jeopardize compliance with the protocol.
9. Evidence of the following infections: active infection including tuberculosis; known HIV infection. that is not well controlled; active or uncontrolled HBV or HCV; or active hepatitis A.
10. Active or prior documented autoimmune or inflammatory disorders.
11. Participants who are candidates for curative therapy.
12. Prior exposure to any immune-mediated therapy.
13. Current or prior use of immunosuppressive medication within 14 days before the first dose of the study intervention is excluded. The following are exceptions to this criterion: a) Intranasal, inhaled, topical steroids, or local steroid injections (eg, intraarticular injection); b) Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication or chemotherapy premedication) or a single dose for palliative purpose (eg, pain control).
14. Participants are ineligible if they have received any anti-cancer therapy within 28 days prior to the first dose of study intervention or within 5 half-lives of the respective agent, whichever is longer..
15. Any concurrent chemotherapy except study intervention, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment.
16. Radiotherapy treatment with a wide field of radiation or to more than 30% of the bone marrow within 4 weeks, prior to the first dose of study intervention.
17. Major surgical procedures within 4 weeks prior to the first dose of the study intervention or still recovering from prior surgery.
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of the study intervention.
19. Participants with a known allergy or hypersensitivity to any study intervention, on any excipients of any study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 3 years
  Confirmed ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR, as determined by Investigator per RECIST 1.1.
The number of participants with adverse events/serious adverse events | Through study completion, an average of 3 years
  Number of participants with adverse events and with serious adverse events including abnormal clinical observations, abnormal Electrocardiogram (ECG) parameters, abnormal laboratory assessments and abnormal vital signs that changed from baseline.

SECONDARY OUTCOMES:
Duration Of Response (DOR) | Through study completion, an average of 3 years
  DoR is defined as the time from the date of first documented confirmed response (which is subsequently confirmed) until date of documented progression per RECIST 1.1 as assessed by Investigator or ICR, or death due to any cause.
Progression free survival (PFS) | Through study completion, an average of 3 years
  PFS is defined as the time from date of first dose of study intervention until progression per RECIST 1.1 as assessed by Investigator or ICR, or death due to any cause.
Time to response (TTR) | Through study completion, an average of 3 years
  TTR is defined as the time from the date of the first dose of study intervention until the date of first documented objective response, which is subsequently confirmed per RECIST 1.1, as assessed by Investigator or ICR.
Overall Survival (OS) | Through study completion, an average of 3 years
  OS is defined as the time from the date of first dose of study intervention until the date of death due to any cause.
PK of volrustomig | Through study completion, an average of 3 years
  Concentration of Volrustomig in serum.
The immunogenicity of volrustomig | Through study completion, an average of 3 years
  Incidence of ADAs against volrustomig in serum.
Disease control rate (DCR) | Through study completion, an average of 3 years
  Disease control rate is defined as the proportion of participants with a BOR of confirmed CR, confirmed PR, or SD, as determined by Investigator per RECIST 1.1.
PFS landmark | Through study completion, an average of 3 years
  The landmark of PFS rates at 6, 9, and 12 months.
OS landmark | Through study completion, an average of 3 years
  The median OS and the landmark of OS rate at 12 months.

CONTACTS AND LOCATIONS:
Locations (33):
- United States (4):
  - Research Site, Los Angeles, California
  - Research Site, Baltimore, Maryland
  - Research Site, Stony Brook, New York
  - Research Site, Columbus, Ohio
- Brazil (4):
  - Research Site, Ijuí
  - Research Site, Londrina
  - Research Site, São Caetano do Sul
  - Research Site, Vitória
- China (19):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongguan
  - Research Site, Fuzhou
  - Research Site, Hangzhou
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Wuhou District
- South Korea (2):
  - Research Site, Namdong-gu
  - Research Site, Seoul
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home